CLINICAL TRIAL: NCT06879392
Title: Examination of Physiotherapists' Knowledge, Awareness and Competence on Physical Activity and Exercise in Hemophilia Patients
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Özge Çoban, Assistant Professor, Saglik Bilimleri Universitesi
Other Study IDs: 2025-79
Record Dates: First submitted 2025-03-08; First posted 2025-03-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia
Keywords: Hemophilia; physical activity; exercise; physiotherapists; knowledge; awareness; sufficiency
MeSH Terms: conditions — Hemophilia A; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- physiotherapists: A physiotherapist is a healthcare professional who uses various techniques and methods to treat, prevent, and improve movement and functional impairments. Physiotherapists help restore the normal function of body systems such as the musculoskeletal, nervous, and cardiopulmonary systems.

SUMMARY:
This study aims to assess physiotherapists' knowledge levels, awareness, perceived roles, adequacy of education received, learning preferences, and external barriers regarding exercise and physical activity in individuals with hemophilia. The findings will help identify physiotherapists' educational needs and contribute to the development of strategies to enhance their effectiveness in hemophilia management.

DETAILED DESCRIPTION:
Hemophilia is a congenital bleeding disorder that leads to intra-articular bleeding and musculoskeletal damage, significantly reducing the quality of life. Although physical activity and physiotherapy play a crucial role in preserving joint health, a lack of knowledge and misconceptions cause patients to avoid exercise. Physiotherapists hold a critical role in this process; however, data on their education and awareness levels remain insufficient. Therefore, identifying the educational needs of physiotherapists and enhancing their capacity to guide patients is of great importance.

Study Objective This study aims to assess the knowledge levels, awareness, perceived roles, and educational adequacy of physiotherapists regarding exercise and physical activity in hemophilia patients. Additionally, it seeks to examine physiotherapists' learning preferences and the external barriers they face, contributing to the development of strategies to address these gaps. The findings will serve as a foundation for improving physiotherapists' ability to provide guidance and education to hemophilia patients.

Study Design and Methodology This research is designed as a cross-sectional, online survey study targeting physiotherapists. The reporting of the survey will be conducted using a checklist developed for internet-based e-surveys.

Survey Development

The survey will be developed by a team of experts, including:

A graduate student in physiotherapy and rehabilitation, Two doctoral-level researchers working as academicians, A hematology specialist with ten years of experience in treating hemophilia patients.

The content of the survey will be based on the guidelines developed by the World Federation of Hemophilia. A mixed-question format (multiple-choice, Likert scales, open-ended questions) will be used.

The survey will cover the following topics:

Knowledge level regarding physical activity and exercise education in hemophilia patients, Perceived role, competence, and external factors affecting exercise prescription, Learning preferences, Participants' years of experience and postgraduate education status. Pilot Study and Data Collection The survey will first be piloted with five physiotherapists within the clinical network. At this stage, minor modifications will be made to improve question clarity if necessary. The final version of the survey will be created using Google Forms and distributed to participants via email and WhatsApp.

The survey's introduction section will include:

Estimated completion time, Data storage methods, Researcher identities, Study objectives, A checkbox for participants to provide informed consent.

Data Analysis In addition to questions assessing knowledge levels, participants' perceptions of their knowledge, education, skills, confidence, and role will be evaluated using a Likert scale (ranging from "strongly agree" to "strongly disagree"). Furthermore, participants' learning preferences and external factors influencing their learning process regarding exercise and physical activity in hemophilia patients will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Profession Group: Participants must be physiotherapists.

Exclusion Criteria:

* Non-Physiotherapists: Individuals who are not licensed physiotherapists will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 300
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Physiotherapists' Knowledge | From March 2025 to June 2025
  One of the primary outcomes of this study is physiotherapists' knowledge level about physical activity and exercise in hemophilia patients.The knowledge level of physiotherapists will be measured with the questionnaire developed.
Physiotherapists' Awareness | From March 2025 to June 2025
  One of the primary outcomes of this study is physiotherapists' awareness level about physical activity and exercise in hemophilia patients.One of the primary outcomes of this study is physiotherapists' knowledge level about physical activity and exercise in hemophilia patients.The wareness level of physiotherapists will be measured with the questionnaire developed.
Physiotherapists' Competence | From March 2025 to June 2025
  One of the primary outcomes of this study is physiotherapists' competence level about physical activity and exercise in hemophilia patients.The competence level of physiotherapists will be measured with the questionnaire developed.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Gülhane Faculty of Physiotherapy and Rehabilitation, Ankara, Keçiören, Turkey (Türkiye)